CLINICAL TRIAL: NCT02017158
Title: Virtual Sprouts: Web-based Gardening Games to Teach Nutrition and Combat Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Donna Spruijt-Metz, Director, USC/CESR Mobile and Connected Health Program, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-11-00158; R25RR032159 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-20 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Obesity; Nutrition; Children
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Sprouts (Experimental): The Virtual Sprouts intervention arm will play Virtual Sprouts in a school-based implementation of the game.
  Interventions: Other: Virtual Sprouts
- Control group (No Intervention): The control group will consist of students who will not play the Virtual Sprouts game at school.

INTERVENTIONS:
Other: Virtual Sprouts — The Virtual Sprouts intervention group will play Virtual Sprouts in a school-based implementation of the game.
  Arms: Virtual Sprouts

SUMMARY:
The purpose of this study is to develop, disseminate, and evaluate a web-based nutrition and gardening game using interactive, multiplatform and mobile gaming, rich narrative, a pedagogical agent, meaningful play, and experiential learning to prevent/treat obesity in minority 3-5th grade youth and their families.

DETAILED DESCRIPTION:
1-16

C.1.a: Overview of the Plan: This project will proceed in three iterative phases: Development, Dissemination and Evaluation. Development of a) curriculum, b) virtual garden and c) pedagogical agent will proceed in parallel, and be integrated during testing and evaluation. A participatory research group comprised of key community members, teachers, clinicians, education experts, 8-11 year old youth and their parents will be formed to provide iterative rounds of input and evaluation throughout the development of Virtual Sprouts. This participatory research group will provide input through focus groups, beta testing, idea-building and advisement throughout the development of Virtual Sprouts. We have successfully used this model in previous health and intervention studies. The participatory research group is composed of about 20 diverse members so as not to tax individual members with study needs and to ensure diverse input. Sub-groups of the larger participatory research group are formed for specific tasks, depending on research needs and group interest. The Virtual Sprouts Game will be developed around a virtual pedagogical agent, who will guide the player through the game using cognitive and affective learning principles. The Virtual Environment will be a game system developed using deep narrative and dramatic elements. Both the pedagogical agent and game environment will be extensively and iteratively tested with members of our participatory research group during development. The Virtual Sprouts game will then be introduced into three of the USC Family of Schools Elementary schools, C.1.b: Curriculum Development: During the first year of this grant, we will work on developing and focus group testing the nutrition and gardening curriculum. Curriculum will be tested iterative through focus groups and beta testing with members of the participatory research group. The gardening and nutrition program will not only teach children about the health benefits of fruits and vegetables but children will learn additional skills in math, science, and history. The program will include lessons relating to culture, including growing crops that have cultural significance such as nopales, beans, corn and squash (the latter three crops are historically referred to as "the three sisters"). Gardening provides an ideal vehicle for teaching Science, Technology, Engineering, and Mathematics (STEM) topics such as how plants grow and how gardens can be managed in an environmentally sound manner (science including biology, earth sciences, agriculture, and the study of weather and climate), how to make good nutrition choices with the produce they harvest (nutrition sciences, health behavior). Furthermore, thinking about planting, harvesting, and climate involves a great deal of math and engineering. The web-based interactive nature of the Virtual Sprouts game will introduce children to new uses for advanced technologies.

C.1.c: Game, Pedagogical Agent and Virtual Environment Integration: The game will contain the Pedagogical Agent and Virtual Environment and will provide the interaction framework through play mechanics. Rather than a serial task-driven game, we envision a persistent virtual environment in which the player will explore Virtual Sprouts and be challenged and nurtured by the agent in joint social play activities. Play experience will be episodic, requiring a few minutes of play per day over several weeks. Certain interactions in the virtual environment will be joint activities (such as watering or harvesting vegetables), and challenges issued by the agent will involve the agent personally. For example, the agent may challenge the learner to plant, grow, and harvest ingredients for a certain recipe, then prepare it. Based on the quality of the learners work, the agent may like or dislike the resulting meal. Use of this kind of intrinsic feedback blurs the line between learning and gameplay, and makes the agent an integral and thus indispensable part of the experience. During the first year, we will determine the breadth (variety) and depth (challenge) of the game experience in relation to gardening and cooking tasks appropriate for the target population through paper prototyping and iterative play testing (Fullerton T, Swain C, Hoffman S., 2008).

C.1.d: Pedagogical Agent Components: The pedagogical agent will consist of several key components that, when combined, provide a knowledgeable, friendly, and entertaining companion for learning in the Virtual Sprouts environment through cognitive-affective approaches. These components include:

1. Expert knowledge: The character will possess of cognitive model of effective gardening and cooking that will allow it to support the activities of the Virtual Sprouts game. This will enable the agent to explain how to create and maintain a healthy garden, harvest and cook items from the garden, and provide explanations of the health benefits of eating organically prepared foods. The expert model will also form the basis for assessment of learner activities to give them credit when they take a correct action (e.g., water at the correct time and amount) and to know when they've made a mistake (e.g., planted two seeds too close to one another). These assessments will feed into the pedagogical decision system.
2. Pedagogical knowledge: The provision of guidance requires a delicate balance of providing timely (and wanted) support while allowing the learner to feel a sense of freedom and remain stay in control to feel a sense of ownership of the garden. Care must therefore be taken in decisions of how and when to provide guidance. Too little guidance can lead to frustration for many users (i.e., the agent should be helpful), while too much may threaten users' feelings of autonomy and freedom in the game environment (i.e., the agent should not be perceived as controlling). Thus, through a combination of unsolicited guidance triggered by evidence of confusion and/or lack of domain knowledge and solicited guidance, when the learner requests help, the agent will seek to be a productive helper while ensuring that the learner is acquiring the needed knowledge and skills to succeed at Virtual Sprouts, and in their regular lives as the relate to eating and exercise.
3. Emotion/affect knowledge: In addition to supporting game play and providing explanations for game events, the agent will also support the learner's affective state. Cultivating and nurturing interest, motivation, and positive feelings about the domain are critical in the pursuit of behavior change, and expressions of empathy from the agent can play into the learner's willingness to remain engaged (McQuiggan, S.W., Rowe, J.P., & Lester, J.C., 2008). These intervention techniques will be implemented in concert with the game- and cognitive-focused tactics described above. For example, a user who is just beginning and has completed his or her first vegetable will receive high praise, which will diminish with time for that specific accomplishment. Similarly, for learners who express a negative perception of gardening and vegetables, the agent will work harder to motivate and entertain.
4. Animation and sound: As discussed above, the appearance of the agent will have an impact on the learner's affective state, both during and after the interaction. A well-known and respected character, such as one modeled after the First Lady (if possible), will increase the chances of establishing familiarity and credibility from the outset. Use of appealing animations and joint activity, such as watering the garden simultaneously, will bolster feelings of co-presence and teamwork. The character's voice, which will be delivered along with subtitles for English as a second language learners, will be chosen based on the preferences of users from the target audience in early testing of the system.

C.1.e: Game, Pedagogical Agent and Virtual Environment Development: The phases of development are outlined below:

1. Domain knowledge and learning objective analysis: (Desurvire, H., & Wiberg, C., 2008).
2. Expert modeling and feedback:
3. Pedagogical agent design & prototyping:
4. Agent and game integration: I
5. Agent visual and content revisions:

C.1.g: Teacher Professional Development: The vehicle for training teachers to use the Virtual Sprout game is a hybrid approach and includes a Summer Teacher Academy (STA) serving as a kick off program with face to case and USC Distance Education Network (DEN) mediated, school site follow-up professional development in elementary school classrooms using a lesson study approach. Teacher academies have been recognized in the teacher education literature as a powerful and impactful way of comprehensively training and supporting teachers (Crowther, D.T., Vilá J.S., Fathman A.K., 2006).

The Summer Teacher Academy: A summer teacher academy (STA) will occur in August each implementation year immediately after year one of the program's development phase and in years 2-5. Through the STA, teachers will be trained annually. The academies will be three days long at USC's campus as each of the target schools are in relative close proximity with USC. Mornings in the academy will be spent learning the nutrition conceptual knowledge, exploring the application and practicing using a guided experiential learning approach to facilitating the game use. The content for the training will be aligned with grades 6-12 California health content standards focused on nutrition and related health. Lesson study, beginning with observational demos and progressing to teacher created role-play will be of focus of the professional development. The teacher participants will spend a portion of the morning observing and practicing Virtual Sprouts game, discussing the application and use of the game in their classrooms. As academic year follow-up, teacher participants will practice using the Virtual Sprouts game application and engage in peer review of game facilitation with fellow teachers (lesson study) in tandem with the USC teacher education experts in their classrooms.

ELIGIBILITY:
Inclusion Criteria:

* Child in 3rd, 4th, or 5th grade

Exclusion Criteria:

* Child in grades earlier than 3rd or later than 5th

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Dietary intake | pre-intervention and post-intervention (approximately 8 weeks apart)
  Change in scores on dietary intake as measured by the Block dietary screener, administered one week pre-intervention and one week post intervention. Length of intervention is approximately six weeks, depending upon how schools schedule the 12 game modules

SECONDARY OUTCOMES:
Preference for fruits and vegetables | Pre-intervention and post-intervention (approximately 8 weeks apart)
  Change in scores on preference for fruit and vegetables as measured by a taste test administered in class one week pre-intervention and one week post intervention. Length of intervention is approximately six weeks, depending upon how schools schedule the 12 game modules
Gardening knowledge | Pre and post intervention (approximately 8 weeks apart)
  Change in scores on gardening knowledge as measured by questionnaire administered one week pre-intervention and one week post intervention. Length of intervention is approximately six weeks, depending upon how schools schedule the 12 game modules

CONTACTS AND LOCATIONS:
Overall Officials: Donna Spruijt-Metz, PhD, Principal Investigator — University of Southern California; Chad Lane, PhD, Principal Investigator — University of Southern California; Giselle Ragusa, PhD, Principal Investigator — University of Southern California; Marientina Gotsis, MFA, Study Director — University of Southern California; Jaimie Davis, PhD, RD, Study Chair — University of Texas at Austin
Locations (2):
- United States (2):
  - Los Angeles Charter Schools, Los Angeles, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twiss J, Dickinson J, Duma S, Kleinman T, Paulsen H, Rilveria L. Community gardens: lessons learned from California Healthy Cities and Communities. Am J Public Health. 2003 Sep;93(9):1435-8. doi: 10.2105/ajph.93.9.1435. PMID 12948958
- [Background] Kipke MD, Iverson E, Moore D, Booker C, Ruelas V, Peters AL, Kaufman F. Food and park environments: neighborhood-level risks for childhood obesity in east Los Angeles. J Adolesc Health. 2007 Apr;40(4):325-33. doi: 10.1016/j.jadohealth.2006.10.021. Epub 2007 Feb 5. PMID 17367725
- [Background] Robinson EJ, Mitchell P. Children's interpretation of messages from a speaker with a false belief. Child Dev. 1992 Jun;63(3):639-52. PMID 1600828